CLINICAL TRIAL: NCT07171775
Title: Clinical and Three-Dimensional Radiographic Assessment of Bioactive Restorative System Following Selective Caries Removal of Deep Lesions: A Two-Year Randomized Controlled Trial
Brief Title: This Study Aims to Clinically Assess and Radiographically Measure the Formed Dentin Bridge Over the Pulp, Utilizing Three-dimensional Imaging Following the Application of a Bioactive Restorative System Versus a Conventional Restorative System After Selective Caries Removal to Soft Dentin Over 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Hamdy Saber Mohamed, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CU-2025-09
Record Dates: First submitted 2025-09-06; First posted 2025-09-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Deep Carious Lesions; Partial Caries Removal; Dentin Bridge
Keywords: deep caries; partial caries removal; selective caries removal; dentin bridge; Bioactive; universal adhesive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a double-blinded trial: participants and outcome assessors/analysts will be blinded to treatment allocation. The operator (E.H.) cannot be blinded due to differences in handling and placement of the two materials
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioactive Restorative System (Experimental): Experimental Group (Bioactive Restorative System):
  Interventions: Procedure: Experimental - Bioactive Restorative System
- Conventional Restorative System (Active Comparator): Control Group (Conventional Restorative System)
  Interventions: Procedure: Active Comparator -Conventional Restorative System

INTERVENTIONS:
Procedure: Experimental - Bioactive Restorative System — Following selective caries removal to soft dentin, the cavity will be restored using a bioactive restorative system consisting of a bioactive universal adhesive followed by placement of a bioactive bulk-fill resin composite.
  Arms: Bioactive Restorative System
Procedure: Active Comparator -Conventional Restorative System — Following selective caries removal to soft dentin, the cavity will be restored using a conventional universal adhesive system followed by placement of a bulk-fill resin composite
  Arms: Conventional Restorative System

SUMMARY:
This clinical trial aims to evaluate dentin bridge formation over the pulp following selective caries removal in permanent teeth with deep carious lesions (ICDAS scores 5-6). A total of 66 patients will be enrolled and randomly allocated to receive either a bioactive restorative system (bioactive universal adhesive combined with a bioactive bulk-fill resin composite) or a conventional non-bioactive restorative system. Clinical assessments, including pulp sensibility testing and patient-reported pain evaluation, together with three-dimensional radiographic analysis using cone beam computed tomography, will be conducted to assess the thickness and quality of reparative dentin bridge formation. Outcomes will be evaluated at baseline and during follow-up periods extending up to 24 months to compare the effectiveness of both restorative approaches in preserving pulp sensibility and promoting dentin-pulp complex repair.

DETAILED DESCRIPTION:
This randomized controlled clinical trial is designed to evaluate the clinical and radiographic outcomes of a bioactive restorative system compared with a conventional restorative system following selective caries removal in permanent molars with deep carious lesions (ICDAS scores 5-6).

A total of 66 eligible patients will be recruited according to predefined inclusion and exclusion criteria and randomly allocated into two parallel groups. After selective removal of carious dentin to soft dentin, cavities will be restored using either a bioactive restorative system (bioactive universal adhesive combined with bioactive bulk-fill resin composite) or a non-bioactive restorative system (conventional universal adhesive and bulk-fill resin composite).

Clinical assessments will include evaluation of pulp sensibility and patient-reported pain, while radiographic assessment of dentin bridge formation-regarding presence, thickness, and quality-will be performed using three-dimensional cone beam computed tomography. Outcomes will be evaluated at baseline and during follow-up periods extending up to 24 months to compare the effectiveness of both restorative approaches in preserving pulp vitality and promoting dentin-pulp complex repair

ELIGIBILITY:
Inclusion Criteria:

Patient-related criteria:

1. Adult patients (age: 18-40 years) of both genders.
2. Good oral hygiene.
3. Willing to sign the informed consent.
4. Cooperative patients who accept the follow-up period.

Tooth-related criteria:

1. Posterior permanent caries (ICDAS 5-6).
2. Radiographically, caries is extending 50% of dentine with a radiopaque layer between the carious lesion and the pulp chamber.
3. Sensitive teeth according to the cold pulp test.
4. Negative response in percussion test.

Exclusion Criteria:

Patient-related criteria:

1. Allergy to any of the restorative materials.
2. Patients undergoing orthodontic treatment with fixed appliances.
3. Pregnant women.
4. Patients with debilitating systemic diseases.
5. Patient who frequently uses analgesics or any drugs that could mask the pain.

Tooth-related criteria:

1. Teeth with previous restorations.
2. Spontaneous pain or prolonged pain (more than 15 s) after the sensitivity test (cold test), which would indicate irreversible pulpitis.
3. Negative sensibility tests, periapical radiolucency, and sensitivity to axial or lateral percussion.
4. Mobile teeth, indicating periodontal disease or trauma.
5. External or internal resorption.
6. Chipped teeth or Cuspal loss

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment of Pulp sensibility. | 24 months
  Thermal pulp test

SECONDARY OUTCOMES:
Clinical assessment of pain. | 24 months
  (Patient-reported outcome measures) by Visual analogue scale The Visual Analogue Scale (VAS) will be used, by which 0 is no pain and 10 is severe pain.
  Pictures will be added to the same, as well as colors to guide the patient during selection of pain severity.
Thickness and quality of Dentin bridge formation | 24 months
  Assess the dentin thickness by using the linear measurement tool and measuring the distance from the base of restoration to the pulp on sagittal, coronal, or cross-sectional images generated from CBCT scans after orientation of the orthogonal planes using the software's vertical and horizontal reference lines

IPD SHARING:
Plan to Share IPD: No